CLINICAL TRIAL: NCT06945120
Title: Efficacy of an Asian Culture-tailored Lung Health (ACT) Intervention on Lung Cancer Screening and Smoking Cessation in Asian Americans
Brief Title: ACT Lung Health Intervention: Phase Two
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Mary E. Cooley, Phd, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 25-041; 5U54CA156734-14 (NIH); 5U54CA156732-14 (NIH)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation; Smoking Behaviors; Smoking, Tobacco; Smoking, Cigarette; Smoking (Tobacco) Addiction
Keywords: Smoking Cessation; Lung Cancer Screening; Smoking (Tobacco) Addiction; Smoking, Cigarette; Smoking, Tobacco; Smoking Behaviors
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Smoking; Cigarette Smoking; Behavior, Addictive | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: ACT Lung Health Intervention (Experimental): Participants will be randomized 1:1 by block size and stratified by ethnicity and readiness to quit smoking and will complete:
  * Baseline visit
  * Questionnaires at 1, 3, and 6 months
  * 3 month saliva test
  * Weekly Zoom sessions
  * 6 month saliva test
  Interventions: Behavioral: ACT Lung Health Intervention
- Group B: Standard Care (No Intervention): Participants will be randomized 1:1 by block size and stratified by ethnicity and readiness to quit smoking and will complete:
  * Baseline visit
  * Questionnaires at 1, 3, and 6 months
  * 3 month saliva test
  * Weekly Zoom sessions
  * 6 month saliva test

INTERVENTIONS:
Behavioral: ACT Lung Health Intervention — An Asian culture-tailored lung health intervention, which includes individual counseling sessions, family coaching, provision of nicotine replacement therapy (NRT) in the form of patches, lozenges, or chewing gum, and educational materials about low-dose computed tomography (LDCT) for lung cancer screening. The eight weekly, counseling sessions with study staff will be conducted via phone call or the Zoom web-conferencing platform.
  Other Names: Asian Culturally Tailored Lung Health (ACT) Intervention
  Arms: Group A: ACT Lung Health Intervention

SUMMARY:
This study aims to test a counseling and educational program designed to improve lung health through smoking cessation for Chinese and Korean American smokers at high risk for lung cancer.

DETAILED DESCRIPTION:
This two-arm stratified randomized clinical trial is to test a counseling and educational program designed to improve lung health through smoking cessation for Chinese and Korean American smokers at high risk for lung cancer.

Participants will be randomized into one of two groups: Group A: ACT Lung Health Intervention versus Group B: Standard Care. Randomization means a participant is placed into a study group by chance.

The research study procedures include screening for eligibility, questionnaires, and saliva tests.

It is expected participation in this study will last about 6 months.

About 60 participants are expected to take part in this research study.

The National Cancer Institute is providing funding for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as either Chinese or Korean
* Speak either Korean, Mandarin, or English
* Eligible for LDCT screening (50-80 years of age and 20- pack-year smoking history)
* Currently smoking (i.e., having smoked within the prior 30 days),
* Currently have active health insurance coverage and a primary healthcare provider and
* Have access to a video-call device with internet or wireless connection.
* Eastern Cooperative Oncology Group functional status <2
* Live in the United States for the next 12 months

Exclusion Criteria:

* Had LDCT screening done within the last 2 years.
* Hospitalization due to a serious mental illness (e.g., psychotic disorders) during the prior 6 months.
* Previous history of lung cancer.
* We will not include any of the following special populations:

  * Adults unable to consent.
  * Adults younger than 50 or older than 80 years
  * Individuals who are not yet adults (infants, children, teenagers)
  * Pregnant women
  * Prisoners

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically Verified 7-Day Point Prevalence Smoking Abstinence at 6 Months (Group A) | 6 months post-baseline assessment
  The proportion of participants who have not smoked cigarettes (not even a puff) in the past 7 days at the 6-month follow-up, verified biochemically using salivary cotinine testing. Participants reporting abstinence and not using nicotine replacement therapy (NRT) will perform a salivary cotinine test observed via video call. Cotinine levels ≤3 ng/mL will confirm abstinence.
Biochemically Verified 7-Day Point Prevalence Smoking Abstinence at 6 Months (Group B) | 6 months post-baseline assessment
  The proportion of participants who have not smoked cigarettes (not even a puff) in the past 7 days at the 6-month follow-up, verified biochemically using salivary cotinine testing. Participants reporting abstinence and not using nicotine replacement therapy (NRT) will perform a salivary cotinine test observed via video call. Cotinine levels ≤3 ng/mL will confirm abstinence.
Completion of Lung Cancer Screening with Low-Dose Computed Tomography (LDCT) at 6 Months (Group A) | Within 6 months post-baseline assessment
  The proportion of participants who have completed lung cancer screening using LDCT within 6 months after baseline assessment. Completion will be verified by self-report and/or by obtaining a copy of the LDCT results from participants.
Completion of Lung Cancer Screening with Low-Dose Computed Tomography (LDCT) at 6 Months (Arm B) | Within 6 months post-baseline assessment
  The proportion of participants who have completed lung cancer screening using LDCT within 6 months after baseline assessment. Completion will be verified by self-report and/or by obtaining a copy of the LDCT results from participants.

SECONDARY OUTCOMES:
Change in Number of Cigarettes Smoked per Day from Baseline to 6 Months (Group A) | Baseline and 6 months post-baseline assessment
  The mean change in the number of cigarettes smoked by participants per day from baseline to 6 months post-baseline.
Change in Number of Cigarettes Smoked per Day from Baseline to 6 Months (Group B) | Baseline and 6 months post-baseline assessment
  The mean change in the number of cigarettes smoked by participants per day from baseline to 6 months post-baseline.
Self-Reported 7-Day Point Prevalence Smoking Abstinence at 3 Months (Group A) | 3 months post-baseline assessment
  The proportion of participants who self-report not smoking cigarettes (not even a puff) in the past 7 days at the 3-month follow-up.
Self-Reported 7-Day Point Prevalence Smoking Abstinence at 3 Months (Group B) | 3 months post-baseline assessment
  The proportion of participants who self-report not smoking cigarettes (not even a puff) in the past 7 days at the 3-month follow-up.
Self-Reported 7-Day Point Prevalence Smoking Abstinence at 6 Months (Group A) | 6 months post-baseline assessment
  The proportion of participants who self-report not smoking cigarettes (not even a puff) in the past 7 days at the 6-month follow-up.
Self-Reported 7-Day Point Prevalence Smoking Abstinence at 6 Months (Group B) | 6 months post-baseline assessment
  The proportion of participants who self-report not smoking cigarettes (not even a puff) in the past 7 days at the 6-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Cooley, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu